CLINICAL TRIAL: NCT02022618
Title: Target Organ Damage and Blood Pressure, Retinal Vessels, Oxidative Stress and Polymorphisms Vav-2 and Vav-3 in Hypertensive Subjects (LOD-Hypertension)
Brief Title: Target Organ Damage and Polymorphisms Vav-2 and Vav-3 in Hypertensive Subjects
Acronym: LOD-HTA
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Other Study IDs: (BIO/SA05/13)
Record Dates: First submitted 2013-12-10; First posted 2013-12-30 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Hypertension; Target organ damage; polymorphism; Hypertensive patients
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human biospecimens used will be collected, stored, used, shared, and disposed of in accordance with the informed consent signed by the subject, or under a waiver of informed consent granted by an independent ethical review body, in accordance to Spanish Law (Ley Orgánica de Protección de Datos de Carácter Personal (15/1999 del 13 de Diciembre, LOPD), y en las condiciones que marca la Ley 14/2007 de investigación biomédica) of Protection of Human Subjects.
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives: To analyze the influence on the presence of target organ damage renal, cardiac and vascular of peripheral and central blood pressure, retinal vessels caliber, oxidative stress and polymorphisms of genes VAV-2-3 in hypertensive subjects.

Methodology: A cross- sectional design we will performed . Population: 486 hypertensive patients. Target organ damage will be assessed by tests recommended in 2013 European guidelines of hypertension. Blood pressure office and ambulatory, retinal caliber vassels,oxidative stress and polymorphisms VAL -2-3 will be measurement.

DETAILED DESCRIPTION:
Ambulatory blood pressure monitoring (ABPM): The ABPM will be performed on a day of standard activity, with an adequate cuff for the size of the patient's arm. A control system, SpaceLabs 90207 model (Spacelabs Healthcare, Issaquah, Washington, USA), validated according to the protocol of the British Hypertension Society, will be used [57]. The records in which the percentage of valid readings will be 80% of the total and with valid readings at all times were considered to be valid. Furthermore, for the records to be evaluable, at least 14 measurements will be required during the daytime period, or at least seven during the nightime or rest period. The monitor will be scheduled for obtaining blood pressure measurements every 20 min during the daytime period and every 30 min during the rest period. The average and dispersion estimators of SBP and DBP were calculated during the 24-h, daytime and nightime periods, defined based on the diary reported by the patient. The patient completes a form specifying bedtime and wake-up time.

Ambulatory arterial stiffness index (AASI) and Home arterial stiffness index (HASI): Arterial stiffness will be evaluated by the ambulatory and home arterial stiffness indices (AASI and HASI). For AASI and HASI estimation, the regression slope of diastolic on systolic blood pressure will be computed for each individual on the basis of 24-hour ABPM (AASI) and also HASI readings over 6 days. AASI as well as HASI were defined as one minus the respective regression slope of DBP on SBP [58]. AASI will also computed from waking or sleeping blood pressure.

Evaluation of retinal vessels: Retinography will be performed using a Topcon TRC NW 200 nonmydriatic retinal camera (Topcon Europe B.C., Capelle a/d Ijssel, The Netherlands), obtaining nasal and temporal images centered on the disk. The nasal image with the centered disk will be loaded into the developed software, AV Index calculator (Ciclorisk SL, Salamanca, Spain, registry no. 00/2011/589). The software automatically recognizes the disk and draws two external concentric circles which delimit area A, between 0 and 0.5 disk diameters from the optic disk margin, and area B, between 0.5 and 1 disk diameters from the margin. The software first identifies the limits of the different vessels, after which it automatically recognizes arteries and veins, and makes multiple measurements of the diameter of the section of the vessels circulating through area B. It finally estimates the mean caliber of veins and arteries in mm, and these measurements are summarized as an arteriole-venule ratio, AVIx. An AVIx of 1.0 suggests that arteriolar diameters will be on average the same as venular diameters in that eye, whereas a smaller AVR suggests narrower arterioles. We used the pairs of main vessels in the upper and lower temporal quadrants, rejecting all other vessels, to improve reliability and increase efficiency of the process, analyzing measures for each quadrant separately and together to estimate the mean measure in each eye. [64].

Laboratory:Determining the concentration of superoxide and catecholamines (adrenaline and noradrenaline) in plasma and urine anion will be determined by ELISA (CatCombi ELISA, IBL, Deventer, The Netherlands), following the manufacturers instructions. Superoxide dismutase activity in plasma will be also assessed using ELISA kits (Cu-Zn superoxid-dismutase ELISA, IBL), and the urinary excretion and plasma levels of lipid peroxides by measuring products react with thiobarbituric acid (TBARS) (OxiSelect TBARS Assay Kit, Cell Biolabs, Inc., San Diego, CA 92126).

In a sample of DNA from peripheral blood erythrocyte polymorphisms of VAV and VAV-2-3 genes in all study subjects are studied. To this end, 10cc of venous blood obtained with anticoagulant (EDTA: ethylene diamine tetra-acetic acid).

Renal assessment: The kidney damage will be assessed by measuring creatinine plasma concentration, the glomerular filtration rate was estimated by CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) [59] and the MDRD-IDMS (Modification of Diet in Renal Disease-Isotopic Dilution Mass Spectrometry) [60] equation and proteinuria were assessed by the albumin/creatinine ratio following the 2007 European Society of Hypertension/European Society of Cardiology Guidelines criteria [2]. Subclinical organ damage was defined as plasma creatinine between 1.3 - 1.5 mg/dl in men and 1.2 - 1.4 mg/dl in women, glomerular filtration rate below 60 ml/min or albumin/creatinine ratio > 22 mg/gr in men and 31 mg/ gr in women. Renal disease was defined as plasma creatinine of 1.5 mg/dl or higher in men and 1.4 mg/l in women or albumin/creatinine ratio > 300 mg/24 h.

Cardiac assessment: The electrocardiographic examination will be performed with a General Electric MAC 3.500 ECG System (Niskayuna, New York, USA), that measures automatically the voltage and duration of waves and estimates the criteria of the Cornell voltage-duration product (Cornell VDP) [61] to assess the LVH by the following equation: Men ((RaVL + SV3) * QRS) and women ((RaVL + SV3) * QRS + 6). LVH will be defined as the voltage-duration product > 2,440 mm/ms [2] and Sokolow and R avl > 11.

Pulse wave velocity (PWV): These parameters will be estimated using the SphygmoCor System (AtCor Medical Pty Ltd., Head Office, West Ryde, Australia). Using the SphygmoCor System (Vx pulse wave velocity), and with the patient in the supine position, the pulse waves of the carotid and femoral arteries were analyzed, estimating the delay with respect to the ECG wave and calculating PWV. Distance measurements were taken with a measuring tape from the sternal notch to the carotid and femoral arteries at the sensor location [62].

Assessment of vascular structure by carotid intima media thickness (IMT): Carotid ultrasound to assess C-IMT will be performed by two investigators trained for this purpose before starting the study. The reliability of such recordings was evaluated before the study, using the intraclass correlation coefficient, which showed values of 0.97 (95%CI: 0.94-0.99) for intra-observer agreement on repeated measurements in 20 subjects, and 0.90 (95%CI: 0.74-0.96) for inter-observer agreement. According to the Bland-Altman analysis, the limit of inter-observer agreement was 0.02 (95% CI: -0.05-0.10), while the limit of intra-observer agreement was 0.01 (95% CI: -0.03-0.06). A Sonosite Micromax ultrasound device paired with a 5-10 MHz multi-frequency high-resolution linear transducer with Sonocal software will be used for performing automatic measurements of carotid IMT in order to optimize reproducibility. Measurements will be made of the common carotid after the examination of a 10-mm longitudinal section at a distance of 1 cm from the bifurcation, performing measurements in the anterior or proximal wall, and in the posterior or distal wall in the lateral, anterior and posterior projections, following an axis perpendicular to the artery to discriminate two lines: one for the intima-blood interface and the other for the media-adventitious interface. A total of 6 measurements will be obtained of the right carotid, with another 6 measurements of the left carotid, using average values (average carotid IMT) and maximum values (maximum carotid IMT) automatically calculated by the software [63]. The measurements will be obtained with the subject lying down, with the head extended and slightly turned opposite to the examined carotid artery. The average IMT will considered abnormal if it measured 0.90 mm, or if there will be atherosclerotic plaques with a diameter of 1.5 mm or a focal increase of 0.5 mm or 50% of the adjacent IMT [2].

ELIGIBILITY:
Inclusion Criteria:

Subjects diagnosed of essential hypertension and age between 20-80 years.

Exclusion Criteria:

Participants who do not sign the consent written informed

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: 486 hypertensive patients (20-80 years) will be assessed with all tests recommended in 2013 European guidelines of hypertension
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Target organ damage cardiovascular | 1 year
  Target organ damage, cardiac (left ventricular hypertrophy), Vascular (Pulse wave velocity and Carotid intima media tickness), and renal (Glomerular filtration low and Microalbuminury)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel A Gomez Marcos, MD, Principal Investigator — Fundacion Infosalud
Locations (1):
- La Alamedilla Health center, Salamanca, Salamanca, Spain

REFERENCES:
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] Lorenz MW, Markus HS, Bots ML, Rosvall M, Sitzer M. Prediction of clinical cardiovascular events with carotid intima-media thickness: a systematic review and meta-analysis. Circulation. 2007 Jan 30;115(4):459-67. doi: 10.1161/CIRCULATIONAHA.106.628875. Epub 2007 Jan 22. PMID 17242284
- [Background] Garcia-Ortiz L, Recio-Rodriguez JI, Parra-Sanchez J, Gonzalez Elena LJ, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Gomez-Marcos MA; Vaso-risk group. A new tool to assess retinal vessel caliber. Reliability and validity of measures and their relationship with cardiovascular risk. J Hypertens. 2012 Apr;30(4):770-7. doi: 10.1097/HJH.0b013e3283506628. PMID 22306849
- [Background] Fraser HI, Dendrou CA, Healy B, Rainbow DB, Howlett S, Smink LJ, Gregory S, Steward CA, Todd JA, Peterson LB, Wicker LS. Nonobese diabetic congenic strain analysis of autoimmune diabetes reveals genetic complexity of the Idd18 locus and identifies Vav3 as a candidate gene. J Immunol. 2010 May 1;184(9):5075-84. doi: 10.4049/jimmunol.0903734. Epub 2010 Apr 2. PMID 20363978
- [Derived] Gomez-Marcos MA, Gonzalez-Sarmiento R, Recio-Rodriguez JI, Agudo-Conde C, Gamella-Pozuelo L, Perretta-Tejedor N, Martinez-Salgado C, Garcia-Ortiz L; Members of the LOD-Hipertension Group. Relationship between target organ damage and blood pressure, retinal vessel calibre, oxidative stress and polymorphisms in VAV-2 and VAV-3 genes in patients with hypertension: a case-control study protocol (LOD-Hipertension). BMJ Open. 2014 Apr 3;4(4):e005112. doi: 10.1136/bmjopen-2014-005112. PMID 24699462